CLINICAL TRIAL: NCT05440903
Title: Examining the Effects of Brief Mindfulness Training on Smoking Quit Attempts
Brief Title: Mindfulness Training for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Matthew Kirkpatrick, Associate Professor of Research, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UP-20-00900
Record Dates: First submitted 2022-06-22; First posted 2022-07-01 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Smoking Cessation
Keywords: Mindfulness; Meditation
MeSH Terms: conditions — Smoking Cessation | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Between-groups study design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The investigators and majority of study staff are blinded. The only individuals who are unblinded to a participant's conditions do not conduct data collection nor interact with participants beyond assigning participants to a condition and explaining the protocol for MT or control app training.
  Participants are aware of their condition, but do not know that the protocol is being measured as the variable of interest, nor that other participants are assigned to different conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Experimental): Participants in the experimental arm are asked to use a mindfulness smartphone application called Headspace. Headspace offers pre-recorded introductory mindfulness meditation audio instructions guided by experienced meditation teachers. Study participants are instructed to voluntarily complete 10 minutes of Headspace twice per day for 14 days, a total recommended dose of 280 minutes. Mindfulness practice begins the day after the baseline interview (i.e., intervention day 1). Participants are encouraged to listen at two separate times each day to support habit formation and to maximize daily exposure with low time burden. As participants have minimal prior experience with mindfulness attributed to the study eligibility criteria, all recommended trainings are at the beginner level. Participants have access to all sessions offered and are not restricted to a particular sequence.
  Interventions: Behavioral: Headspace
- Psychoeducation (Placebo Comparator): Participants in the psychoeducation arm listen to TEDTalks audio recordings by experts on field-specific topics. Study participants are instructed to complete 10 minutes of TEDTalks twice per day for 14 days. Sessions were selected by the study team to be of interest to the public yet not include content on meditation, smoking, or content appearing to cue behavior change associated with smoking. Like the Mindfulness condition, participants in the Psychoeducation condition begin the practice the day after the baseline interview. Participants are told to listen at two separate times each day to maximize daily exposure with low time burden. Additionally, participants are instructed to listen with "full mindful attention and return attention to the audio when attention drifts" to match the Mindfulness instruction and emphasize the importance of sustaining attention for each 10-minute period. Participants have access to all sessions offered and are not restricted to a particular sequence.
  Interventions: Behavioral: TEDTalk

INTERVENTIONS:
Behavioral: Headspace — A smartphone application that provides users with mindfulness and meditation sessions.
  Other Names: Mindfulness
  Arms: Mindfulness
Behavioral: TEDTalk — A smartphone application that provides users with psychoeducational audio recordings from TEDTalk.
  Arms: Psychoeducation

SUMMARY:
Participants will complete this study remotely, either at home or at their preferred location using an online platform. The investigators propose to test the effects of a mindfulness training [MT: Headspace] intervention compared to a time and attention psycho-education control [control: TedTalks] among N=200 adult smokers of a nicotine product. Previous studies suggest that mindfulness training may be beneficial in reducing craving during tobacco abstinence. During the study, participants will complete baseline questionnaires, followed by two weeks of daily MT or control training and self-report on questionnaires assessing affect, cognition, and smoking behavior using Ecological Momentary Assessment (EMA) for remote data capture. Following this two weeks of training, participants will complete a smoking quit attempt and complete daily EMA questionnaires for two weeks. The first day of the smoking quit attempt will include a remote Zoom video session following overnight smoking abstinence. During this session the participants will complete a remote stressor task (Trier Social Stress Test, TSST), and the investigators will collect EMA data on affect and smoking behavior before and after the TSST. One month after the start of the quit attempt, participants will complete a phone call as a follow-up to assess smoking behavior over the previous 30 days, and to complete a debriefing. Study objectives are to test the effect of MT on: (1) smoking lapses during the follow-up periods; and (2) stress (affect, smoking urge, withdrawal symptoms) during the TSST.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Smoke at least 5 cig/day for the past year
* English fluency
* Motivation to quit smoking in next 30 days, or willing to make a practice quit attempt
* Reside in California
* Have remote video capability (i.e., computer, laptop, tablet with working camera and audio) in order to complete all data collection procedures (Note that the study does not have resources to provide these materials)
* Have working smartphone capable of downloading the app for EMA assessments

Exclusion Criteria:

* Current use of any nicotine replacement products (i.e., nicotine patch, gum, lozenge) or smoking cessation medications (i.e., Chantix, Bupropion, Wellbutrin, Zyban)
* Current mindfulness or meditation practice of greater than 5 minutes each day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Smoking Cessation Behavior at 14 days | 14 days after start of quit attempt
  7-day point prevalence abstinence (i.e., no cigarettes smoked in the previous 7 days). 0=did not smoke; 1=smoked at least one cigarette.
Smoking Cessation Behavior at 30 days | 30 days after start of quit attempt
  7-day point prevalence abstinence (i.e., no cigarettes smoked in the previous 7 days). 0=did not smoke; 1=smoked at least one cigarette.

SECONDARY OUTCOMES:
Cessation Motivation | baseline (start of the study) and 30 days after start of quit attempt
  change in motivation to quit (or stay quit) as measured by the Contemplation Ladder, a visual graphic used to select current level of quit motivation (0="no thought of quitting"; 10="taking action to quit"). A higher number indicates greater motivation to quit smoking.
App training adherence | 14 days after starting app training
  Adherence to app use will be calculated as the number of times an individual used the app out of a total of 28 sessions (2 session per day for 14 days). A higher number indicates better adherence.
Stress-related feelings of "anxious" | 1 min before the Trier Social Stress Test (TSST), and +5, +30, +60 min after TSST
  visual analog scales of "I feel anxious" using the scale (0="not at all" to 100="extremely"). A higher number indicates greater feelings of "anxious"
Stress-related feelings of "relaxed" | 1 min before the Trier Social Stress Test (TSST), and +5, +30, +60 min after TSST
  visual analog scales of "I feel relaxed" using the scale (0="not at all" to 100="extremely"). A higher number indicates greater feelings of "relaxed"
Stress-related feelings of "stressed" | 1 min before the Trier Social Stress Test (TSST), and +5, +30, +60 min after TSST
  visual analog scales of "I feel stressed" using the scale (0="not at all" to 100="extremely"). A higher number indicates greater feelings of "stressed"
Stress-related feelings of "urge to smoke" | 1 min before the Trier Social Stress Test (TSST), and +5, +30, +60 min after TSST
  visual analog scales of "I have an urge to smoke" using the scale (0="not at all" to 100="extremely"). A higher number indicates greater feelings of "urge to smoke"

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Kirkpatrick, Ph.D., Principal Investigator — Associate Professor of Research
Locations (1):
- Keck School of Medicine of USC, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan on sharing deidentified data with other researchers by request.

REFERENCES:
- [Derived] Black DS, Kirkpatrick M. Test of daily app-based mindfulness meditation preceding a planned smoking quit attempt date on abstinence: Protocol for a randomized controlled trial recruiting across the 58 counties of California. Contemp Clin Trials. 2022 Sep;120:106855. doi: 10.1016/j.cct.2022.106855. Epub 2022 Jul 18. PMID 35863695